CLINICAL TRIAL: NCT00194181
Title: Randomized Prospective Trial of Rt-PA Infusion Versus Catheter Exchange for Treatment of Dialysis Catheter Malfunction Due to Fibrin Sheath Formation
Brief Title: Rt-PA Infusion Versus Catheter Exchange for Dialysis Catheter Malfunction Due to Fibrin Sheath
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 705565
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-07-17 (Estimated); Status verified 2006-07

CONDITIONS: Dialysis Catheter Fibrin Sheath; Clotted Dialysis Catheter; Catheter Malfunction
Keywords: dialysis; fibrin; sheath; clot; tpa

INTERVENTIONS:
Drug: TPA Infusion

SUMMARY:
Treating central venous dialysis catheter malfunction due to fibrin sheath formation with rt-PA(TPA)infusion will give equal patency rates in a more cost effective manner when compared to catheter exchange.

Subjects are randomized to TPA infusion or catheter exchange and then followed for catheter function at the post treatment dialysis session, 30-day dialysis session and 60-day dialysis session. Costs and treatment results will be compared.

DETAILED DESCRIPTION:
Patients who come to the Hospital of the University of Pennsylvania, Presbyterian Medical Center or American Access in Northeast Philadelphia with a dialysis catheter that's not functioning well, will be screened for this study.

If the patient qualifies and consents to participate, an envelope will be opened that tells us to exchange the catheter for a new one OR infuse TPA (clot-dissolving drug) into the 2 ports for two and a half hours. Some dialysis patients have had a TPA "dwell" at the dialysis clinic to help increase blood flow during dialysis. The motion of the "infusion" of TPA is expected to be more effective than a "dwell" that sits still. Also, there is more TPA used during "infusion" than during the "dwell".

Once the catheter is functioning, the patient goes home as usual and follow-up is done by phone after the next dialysis session, at 30 days and at 60 days. Follow-up is done to check for flow rates during dialysis and to check for any problems related to the catheter treatment. Participation is complete after the 60-day follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tunneled hemodialysis catheters who have clinical evidence of catheter tip clot and fibrin sheath formation

Exclusion Criteria:

* Malpositioned or kinked catheter requiring catheter change
* Complete thrombosis of the catheterized vein
* Evidence of catheter related infection
* GI bleed within 6 weeks
* Cerebral Infarct within 6 months
* Major surgery within 4 weeks
* Platelet count below 25000
* INR above 2.0
* Sepsis
* Pregnancy
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-03; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: S. William Stavropoulos, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States